CLINICAL TRIAL: NCT05900960
Title: Hot or Cold Beverages in Warm Weather: A Double-blinded Randomized Controlled Trial.
Brief Title: Hot or Cold Beverages in Warm Weather
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Siv Fonnes, Doctor, Herlev Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: F-23023485
Record Dates: First submitted 2023-04-27; First posted 2023-06-13 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Quality of Life
MeSH Terms: interventions — Tea

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Warm tea (Experimental): 50 degrees celsius hot tea.
  Interventions: Dietary Supplement: Tea
- Cool tea (Active Comparator): 10 degrees celsius cool tea
  Interventions: Dietary Supplement: Tea

INTERVENTIONS:
Dietary Supplement: Tea — Orally administered. Decaffeinated tea, with no additives (sugar, honey, etc.)

SUMMARY:
Some studies have suggested that hot beverages are better for cooling down when body temperature rises. No study has investigated the effect of hot beverages in hot weather on personal well-being compared to cold beverages.

DETAILED DESCRIPTION:
The research project will be conducted as a double-blinded randomized crossover trial, where the participants will drink either 10 cl of 10°C cold tea (±2°C) or 50°C hot tea (±2°C), which in a pilot study and in the literature [1,9] has been shown to be without discomfort or side effects. The order of the two interventions will be randomized.

All participants must be adults (18 years or older) and not have a fever on the day of the experiment.

Prior to participation, participants must provide written informed consent and must show up in clothing they find comfortable in the sun and be wearing sunscreen and a sun hat/cap. Participants must also complete a questionnaire on basic background information: gender, age, height, weight, clothing during the trial, and the participant's preference regarding the climate and temperature of beverages.

Walk-through of study:

1. Participants lie or sit in the sun for 10 minutes without drinking anything.
2. Then, participants drink their allocated beverage in ≤ 5 sec. while still in the sun.
3. Approximately 3 minutes (±1 min.) after ingestion of the beverage intervention, participants must answer all questionnaires and have their temperature measured.
4. Afterward, participants stay in the shade for 5 minutes (wash-out period).
5. Participants lie down (or sit) in the sun for the second time for 10 minutes without drinking anything.
6. Then, participants drink their second allocated beverage in ≤ 5 sec. while still in the sun.
7. Approximately 3 minutes (±1 min.) after ingestion of the second beverage intervention, participants must again answer all questionnaires and have their temperature measured.
8. Data collection and the research project end thereafter

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Must be able to ingest intervention
* Must be able to be in the sun for 2x 13 minutes (using sunscreen and/or other relevant UV protection).

Exclusion Criteria:

* Fever on the day of the experiment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-05-09 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2023-05-10 (Actual)

PRIMARY OUTCOMES:
Thermal well-being | At 3 minutes after intervention
  Using the Bedford thermal comfort scale and ASHRAE thermal sensation scale (-3 to 3, higher is hotter)
Mood | At 3 minutes after intervention
  Using the Brief Mood Introspection Scale (-24 to 24, higher is more positive)
Pain, discomfort, depression. | At 3 minutes after intervention
  Using the 5th domain of the EQ-5D-5L (1-5, higher is more pain and/or discomfort, and more depressed)

SECONDARY OUTCOMES:
Temperature | At 3 minutes after intervention
  Using a forehead thermometer in degrees celsius

CONTACTS AND LOCATIONS:
Overall Officials: Viktor FB Moseholm, Principal Investigator — University of Copenhagen, Herlev Hospital; Jacob Rosenberg, Professor, Study Chair — University of Copenhagen, Herlev Hospital
Locations (1):
- Conference hotel, Kusadasi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moseholm VB, Reistrup H, Rosenberg J, Fonnes S. Christmas article: Well-being in hot weather - a randomised crossover trial. Ugeskr Laeger. 2023 Dec 11;185(50):V20239. Danish. PMID 38084617